CLINICAL TRIAL: NCT06846489
Title: Acalabrutinib Plus Rituximab for the Treatment of Elderly or Low- to Intermediate-Risk Younger Untreated Mantle Cell Lymphoma: A Single-Arm, Open-Label, Multicenter, Phase II Study
Brief Title: Acalabrutinib Plus Rituximab for the Treatment of Elderly or Low- to Intermediate-Risk Younger Untreated Mantle Cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Qingqing Cai, MD. PhD., Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2024-843
Record Dates: First submitted 2025-02-16; First posted 2025-02-26 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-02

CONDITIONS: Mantle Cell Lymphoma (MCL)
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — acalabrutinib; Rituximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acalabrutinib in combination with Rituximab (Experimental): Eligible patients will receive:
  Acalbrutinib : 100 mg bid po, continue treatment until disease progression, intolerable toxicity, or completion of 24 months of treatment.
  Rituximab: 375 mg/m² IV, once weekly during the first cycle, then once monthly for 12 months, followed by once every 2 months, for a maximum of 24 months.
  Interventions: Drug: Acalabrutinib; Drug: Rituximab

INTERVENTIONS:
Drug: Acalabrutinib — 100 mg bid po, continue treatment until disease progression, intolerable toxicity, or completion of 24 months of treatment.
Drug: Rituximab — 375 mg/m² IV, once weekly during the first cycle, then once monthly for 12 months, followed by once every 2 months, for a maximum of 24 months

SUMMARY:
This is a single- arm, open-label, multicenter, phase II study to evaluate Acalabrutinib plus Rituximab for the treatment of elderly or low- to intermediate-risk younger untreated mantle cell lymphoma

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy and safety of Acalabrutinib plus Rituximab for the treatment of elderly or low- to intermediate-risk younger untreated mantle cell lymphoma

Treatrment:

1. Acalabrutinib: 100 mg bid po, continue treatment until disease progression, intolerable toxicity, or completion of 24 months of treatment
2. Rituximab: 375 mg/m2 IV, once weekly during the first cycle, then once monthly for 12 months, followed by once every 2 months, for a maximum of 24 months.

The primary study endpoint is the investigator-assessed complete response (CR) rate at 12 months.

ELIGIBILITY:
Key inclusion Criteria:

1. Age ≥18 years.
2. Histologically confirmed CD20+ mantle cell lymphoma.
3. No prior anti-lymphoma treatment.
4. Ann Arbor stage II-IV.
5. ECOG performance status 0-2, no deterioration >2 weeks before baseline or first dose.
6. Younger subjects (<65) must meet:

   1. Low to intermediate risk sMIPI (0-5)
   2. Ki67 < 50%
   3. No TP53 mutation (NGS)
   4. Lesion diameter ≤5 cm
   5. Non-blastoid, polymorphic disease
7. At least one assessable lesion per Lugano 2014 criteria.
8. Adequate organ and bone marrow function during screening.
9. Female subjects must use contraception as per local regulations.
10. Male subjects must agree to avoid sperm donation during the study and for 12 months post-rituximab.
11. Willing to undergo all required assessments and procedures, including swallowing capsules/tablets.
12. Able to understand the study's purpose and risks, and provide signed informed consent with authorization for the use of personal health information.

Key exclusion Criteria:

1. Participants with tumor burden reduction prior to stem cell transplantation.
2. History of active lymphoma central nervous system (CNS) involvement, leptomeningeal disease, or spinal cord compression.
3. Any disease evidence deemed by the investigator to be detrimental to the patient's participation or likely to affect protocol adherence (e.g., severe or uncontrolled systemic disease, including uncontrolled hypertension or kidney transplant).
4. History of progressive multifocal leukoencephalopathy (PML) or current diagnosis of PML.
5. Received any investigational drug within 30 days (or 5 half-lives, whichever is shorter) prior to the first dose of the investigational drug.
6. Underwent major surgery within 30 days prior to the first dose of the investigational drug. Note: If the participant has undergone major surgery, they must be fully recovered from any toxicity and/or complications related to the surgery before the first dose.
7. A history of malignancy that could affect protocol adherence or interpretation of results, except for: a. Basal cell carcinoma, squamous cell carcinoma of the skin, cervical carcinoma in situ, or prostate carcinoma in situ treated curatively at any time before the study. b. Other cancers that were treated surgically and/or with radiation, with no disease for ≥3 years without further treatment.
8. Significant cardiovascular disease, such as symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months before screening, or any NYHA Class 3 or 4 heart disease during screening. Note:Participants with well-controlled, asymptomatic atrial fibrillation are allowed.
9. Refractory nausea and vomiting, difficulty swallowing formulations, or malabsorption syndrome; chronic gastrointestinal disease, gastric bypass, or weight-loss surgery (e.g., Roux-en-Y); partial or complete bowel obstruction, or previous major intestinal surgery that may interfere with the absorption, distribution, metabolism, or elimination of the investigational drug.
10. Received a live-virus vaccine within 28 days prior to the first dose of the investigational drug.
11. Known HIV infection.
12. Any active major infection (e.g., bacterial, viral, or fungal, including subjects with positive CMV DNA PCR).
13. Serologic evidence of active hepatitis B or C infection.
14. History of stroke or intracranial hemorrhage within 6 months prior to the first dose of the investigational drug.
15. History of bleeding disorders (e.g., hemophilia, Von Willebrand disease).
16. Requires or is receiving anticoagulation therapy with warfarin or equivalent vitamin K antagonists.
17. Requires strong CYP3A inhibitors or inducers. The use of strong CYP3A inhibitors within 1 week or strong CYP3A inducers within 3 weeks before the first dose of the investigational drug is prohibited.
18. Pregnancy or breastfeeding.
19. Participation in another therapeutic clinical trial.
20. Requires proton pump inhibitor therapy (e.g., omeprazole, esomeprazole, lansoprazole, dexlansoprazole, rabeprazole, or pantoprazole).
21. Currently has a life-threatening disease, medical condition, or organ system dysfunction that, in the investigator's judgment, may compromise the participant's safety or place the study at risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2033-02-10 (Estimated); Study Completion 2033-02-20 (Estimated)

PRIMARY OUTCOMES:
Complete Response(CR) | From the start of treatment with the investigational drug until 12 months
  Defined as the proportion of patients who achieve complete remission

SECONDARY OUTCOMES:
Objective response rate(ORR) | From the start of treatment with the investigational drug until 12 months
  The proportion of patients who achieve complete remission (CR) or partial remission (PR) .
Duration of Response(DOR) | The time from the patient's first efficacy assessment achieving CR or PR until disease progression, up to 5 years
  To investigate the preliminary anti-tumor efficacy
Progression-free survival(PFS) | From the date of enrollment until the date of the first documented progression or date of death from any cause, whichever came first, up to 5 years
  To investigate the preliminary anti-tumor efficacy
Overall survival(OS) | From the date of enrollment until the date of death from ant cause, up to 5 years
  To investigate the preliminary anti-tumor efficacy

CONTACTS AND LOCATIONS:
Locations (1):
- Sun yat-sen university cancer center, Sun yat-sen university, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided